CLINICAL TRIAL: NCT05543551
Title: Effects of Diaphragmatic Breathing With and Without Resistance Program on Functional Capacity and Activity of Daily Living in Post Covid Patients.
Brief Title: Effects of Diagrammatic Breathing With and Without Resistance in Post Covid Patients on ADLs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/0331 Ushma Zulifqar
Record Dates: First submitted 2022-09-15; First posted 2022-09-16 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: COVID-19 Pandemic
Keywords: : COVID, Exercise training, Functional Capacity.
MeSH Terms: conditions — COVID-19 | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diaphragmatic breathing with Resistance Training (Experimental): Diaphragmatic breathing with Resistance Training:
  Wall press-up: Attempt 3 sets of 5 to 10 repetitions. Dumbbell biceps curls: Attempt 3 sets of 5 to 10 repetitions. Back squats: 1 set of 10 repetitions Leg press:1 set of 10 repetitions
  Interventions: Other: Diaphragmatic breathing with Resistance Training
- Diaphragmatic breathing exercises without Resistance Training (Active Comparator): Diaphragmatic Breathing:
  1. Lie on your back on a flat surface (or in bed) with your knees bent. You can use a pillow under your head and your knees for support if that's more comfortable.
  2. Place one hand on your upper chest and the other on your belly, just below your rib cage.
  3. Breathe in slowly through your nose, letting the air in deeply, towards your lower belly. The hand on your chest should remain still, while the one on your belly should rise.
  4. Tighten your abdominal muscles and let them fall inward as you exhale through pursed lips. The hand on your belly should move down to its original position. You can also practice this sitting in a chair, with your knees bent and your shoulders, head, and neck relaxed
  Interventions: Other: diaphragmatic breathing with out resistance training

INTERVENTIONS:
Other: Diaphragmatic breathing with Resistance Training — Wall press-up:
  Stand arm's length from the wall. Place your hands flat against the wall at chest level, with your fingers pointing upwards. With your back straight, slowly bend your arms, keeping your elbows by your side.
  Dumbbell biceps curls:
  Hold a pair of light weights and stand with your feet hip-width. Keeping your arms by your side, slowly bend them until the weight in your hand reaches your shoulder. Slowly lower again.
  Back squats:
  Place barbell with weights onto the squat rack. Bring your body under the bar. Rest barbell over your traps and shoulders. Make sure hands are even on each side of the bar. Keep your feet in the same position as they would be for an air squat. Brace your midline and keep your chest up.
  Leg press:
  Position feet about shoulder width apart. Try to push through your heels, keeping the knees lined up over the toes. Extend the legs until nearly straight, avoiding locking the knees.
  Arms: Diaphragmatic breathing with Resistance Training
Other: diaphragmatic breathing with out resistance training — Diaphragmatic Breathing:
  1. Lie on your back on a flat surface (or in bed) with your knees bent. You can use a pillow under your head and your knees for support if that's more comfortable.
  2. Place one hand on your upper chest and the other on your belly, just below your rib cage.
  3. Breathe in slowly through your nose, letting the air in deeply, towards your lower belly. The hand on your chest should remain still, while the one on your belly should rise.
  4. Tighten your abdominal muscles and let them fall inward as you exhale through pursed lips. The hand on your belly should move down to its original position. You can also practice this sitting in a chair, with your knees bent and your shoulders, head, and neck relaxed
  Arms: Diaphragmatic breathing exercises without Resistance Training

SUMMARY:
Effects of diaphragmatic breathing exercise with and without resistance exercise program on functional capacity and activity of daily living in post covid patients

DETAILED DESCRIPTION:
The pandemic caused by the spread of the COVID-19 virus has implied a major challenge for the health systems and economies all around the world, as well as for their justice institutions; After COVID recovery subject feels muscle weakness and joint stiffness; extreme tiredness (fatigue) and a lack of energy; sleep problems. And these factors disturb the individuals daily activities of life like unable do household chores and social activities. Breathing is a natural process that usually occurs without conscious effort. However, the average breath tends be shallow and does not engage the diaphragm very much. During diaphragmatic breathing, a person consciously engages their diaphragm in order take deeper breaths. A person will notice their stomach rising and falling. They will also feel an expanding or stretching sensation in the stomach, rather than solely in their chest and shoulders. In this research determine the effects of diaphragmatic breathing with and without resistance exercise program on functional capacity and activity of daily living in post COVID patients.

This study will be a randomized controlled trial. This study will be conducted in general hospital Lahore. In the present study under considerations we mainly look on the subjects meeting predetermined inclusion and exclusion criteria will be divided into two groups using lottery method. Sample size will be 42 including both male and female. QUESTIONNAIRE used as subjective measurements and BARTHEL INDEX as objective measurement. PCFS will be used to check the functional capacity and ordinal scale used to measure performance in activities of daily living will be used check activity of daily living. Subjects of one group will be treated with resistance training at both limbs, at upper limb wall press-up and dumbbell biceps curls will be used but at lower limb back squats and leg press will be used and the other group will be treated without resistance training. Each group performed special trainings for 12 weeks, 2 sessions per week; each session took about 1 hour. Protocols were started with 1 set of 10 repetitions at starting baseline and by improving performance and patients' compatibility with trainings, all eventually finished with 3 sets of 20 repetitions at the end of the protocol. Post treatment reading of PCFS and Barthel quality of life will be recorded after every week. Outcome variables will be PCFS, ordinal scale used to measure performance in activities of daily living and pulse oximeter. Data will be analyzed on SPSS-25.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed patients of COVID-19
* patients having age 30 to 60 years of both male and female
* patients who have distributed ADLs due to COVID
* Absence of fever and improvement in respiratory symptoms
* patients who will be willing to participants in the study

Exclusion Criteria:

* any malignant or chronic diseases
* pregnant or lactating women
* poor quality CMR(cardiac magnetic resonance)post recovery
* patients having less than 20 and greater than 60

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2022-09-02 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
Post Covid Functional Status (PCFS): | 8 weeks
  A questionnaire covering the entire range of functional limitations, including changes in lifestyle, sports, and social activities. It was graded as Grade 0, if there was a negligible effect on activities for patients was considered Grade 1, whereas a lower intensity of the activities was considered as Grade 2. Grade 3 accounted for the inability to perform certain accomplishments, forcing patients to structurally modify these. Finally, Grade 4 was reserved for those patients with unembellished functional restrictions.
Barthel Index for Activity of daily living | 8 weeks
  The Barthel Index (BI) measures the extent to which somebody can function independently and has mobility in their activities of daily living feeding, bathing, grooming, dressing, bowel control, bladder control, toileting, chair transfer, ambulation and stair climbing.
Pulse Oximetry | 8 weeks
  Pulse oximeter that measures the proportion of oxygenated hemoglobin in the blood in pulsating vessels, especially the capillaries of the finger or ear.

CONTACTS AND LOCATIONS:
Overall Officials: sumera abdulhameed, MS, Principal Investigator — Riphah International University
Locations (1):
- Iettefaq hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No